CLINICAL TRIAL: NCT01805947
Title: Process-outcome-study in the Context of a Lifestyle Modification Program for Patients With Chronic Pain Conditions
Brief Title: Lifestyle Modification Program for Patients With Chronic Pain Conditions
Acronym: POSITAG
Status: Completed | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principal Investigator, Universität Duisburg-Essen
Other Study IDs: 12-5216 POSITAG
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle Modification: All patients with chronic pain conditions participate in a 8-weeks structured group program. Detailed information on the mindfulness based program can be found in the publication by Paul, A. et al. "An Integrative Day Care Clinic for chronically ill patients: Concept and case presentation" in the European Journal of Integrative Medicine, 2012, 4(4):e455-e459.
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Behavioral: Lifestyle Modification — Lifestyle Modification
  Other Names: see Paul, A. et al.,Eur J Integr Med 2012, 4(4):e455-e459.

SUMMARY:
In this observational study the effects of a Lifestyle Modification Program - offered as a semi-residential day care clinic - on pain, disability, quality of life and satisfaction with life will be investigated. Furthermore the influence of mindfulness, acceptance and coping, and acquired changes in lifestyle behaviors on the outcome after the program will be evaluated.

Effects will be measured after completion of the program (3 months), and at 6 and 12 months follow up after start of the program, i.e. each outcome measure will be taken 4 times within 12 months.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* 18-78
* diagnosed with any chronic pain condition
* physical and mental ability to participate in the program and the study
* written informed consent

Exclusion Criteria:

* participation in any other clinical study focusing on psychological or behavioral intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with pain condition admitted to the lifestyle modification program
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  Pain intensity according to the German Pain Questionnaire (DSF) (Pfingsten et al., 2007), visual analogue scales
Pain intensity | 6 months
  Pain intensity according to the German Pain Questionnaire (DSF) (Pfingsten et al., 2007), visual analogue scales
Pain intensity | 12 months
  Pain intensity according to the German Pain Questionnaire (DSF) (Pfingsten et al., 2007), visual analogue scales

SECONDARY OUTCOMES:
Disability | 3 months
  pain related disability in the domains everyday activity, leisure and work time, visual analogue scales
Disability (PDI) | 3 months
  Pain Disability Index (Dillmann et al., 1994) validated questionnaire
Quality of life (SF-36) | 3 months
  Short Form (36) Health Survey (SF-36) [Bullinger & Kirchberger, 1998].
Depression (BDI) | 3 months
  Beck Depression Inventory (BDI) [Beck, 1987; Hautzinger, 1992]
Life satisfaction (BMLSS) | 3 months
  Brief Multidimensional Life Satisfaction Scale (BMLSS) [Büssing & Fischer, 2009]
Acceptance (ERDA) | 3 months
  Emotional/Rational Disease Acceptance Questionnaire [Büssing et al., 2008, 2010]
Self efficacy | 3 months
  Questionnaire for pain specific self efficacy (FESS) [Mangels et al., 2009)
Coping (AKU) | 3 months
  Questionnaire for adaptive coping (AKU) [Büssing & Fischer, 2009]
Mindfulness (CPSC) | 3 months
  modified Freiburger Mindfulness Inventory (Büssing et al.)
Perceived Stress (PSS-10) | 3 months
  Perceived Stress Scale (PSS-10) [Büssing, 2011)
Inner Congruence (ICPH) | 3 months
  Inner Congruence with the exercise practise of meditation/relaxation/yoga ... (Büssing et al., 2011)
Practice Diary | 3 months
  Patients fill in a week long diary. Measured are the frequency of health behaviors
Experiences with the program | 3 months
  - satisfaction with the program and perceived benefit
Safety of the program | 3 months
  - safety

OTHER OUTCOMES:
Ability and will to change | 3 months
  Ability and will to change (Büssing, 2008)
  - also evaluated at 6 and 12 months
Body awareness (BAQ) | 3 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Body Awareness Questionnaire (BAQ) (Shields 1989)
Body awareness (BRS) | 3 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Body Responsiveness Scale (BRS)(Daubenmier 2005)
Body awareness (SBC) | 3 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Scale of Body Connection (SBC)(Price and Thompson 2007)
Body awareness (PAS) | 3 months
  Newly developed body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Postural Awareness Scale (PAS) (Cramer et al.)
Body awareness (DKB) | 3 months
  The DKB will be used for mediation and moderator analysis with the outcomes and for validation purposes.
  - Dresdner Körperbildfragebogen (DKB)(Pöhlmann et al., 2007)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav J Dobos, Prof, MD, Study Director — University of Duisburg-Essen, Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine; Romy Lauche, PhD, Principal Investigator — University of Duisburg-Essen, Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine; Holger Cramer, PhD, Principal Investigator — University of Duisburg-Essen, Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany